CLINICAL TRIAL: NCT05552612
Title: Quality-of-life in Patients With Long COVID: Harnessing the Scale of Big Data to Quantify the Health and Economic Costs
Brief Title: Health-related Quality of Life and Long COVID
Acronym: OpenPROMPT
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Emily Herrett, Co-Principal Investigator, London School of Hygiene and Tropical Medicine
Other Study IDs: 2022-KEP-799
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long COVID: Patients with Long COVID
- Without Long COVID: Patients who do not have Long COVID

SUMMARY:
Background: Long COVID is estimated to affect 1.7 million people in the UK. One way of assessing the impact of long COVID is to measure quality-of-life through a standard questionnaire, which can then be used to understand the costs of long COVID to the NHS and wider economy. The impact of long COVID on these measures is not currently known. It is important to understand who is worst affected by long COVID and the cost to the National Health Service (NHS), so that strategies like booster vaccines can be prioritised to the right people.

Aim: OpenPROMPT aims to understand the impact of long COVID on quality-of-life in adults in English primary care.

Methods: We will ask people to participate in the study by downloading a smartphone app, and completing a series of questionnaires held within the app. Questionnaires will ask about quality of life, productivity and symptoms of long COVID. Participants will be asked to fill in the questionnaires once a month, for four months. Electronic reminders will be sent to participants to ask them to complete the questionnaires, which will take roughly 15 minutes to complete each month. Participants will also be asked to give consent for linkage of their questionnaire responses to their existing health records.

The results will tell us if long COVID has different quality-of-life and economic impacts among people of different ages, ethnicities, geographic regions, or because of any underlying health conditions. These results can be converted into standardised measurements used by the NHS to measure the impact of illnesses and the cost of long COVID to health services.

Impact: Together with other researchers studying long COVID, we will provide results to support long-term care, and make recommendations for prevention of long COVID in the future. At all stages we will ensure that the input of patients and the public is central to running the study and interpreting the outputs.

Funding: OpenPROMPT is a collaboration between the London School of Hygiene and Tropical Medicine, the OpenSAFELY patient data platform at the University of Oxford, and TPP (which supplies clinical software to General Practices (GPs) in the UK). The project is funded by the National Institute for Health Research.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are that the patient is aged 18 or over and can read and understand English, and can download and use the Airmid app.

Exclusion Criteria:

* The following patients will be excluded:
* Patients under 18 years old;
* Patients who do not have a smartphone or cannot download or log in to the Airmid app;
* Patients who cannot understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who live in England
Sampling Method: Non-Probability Sample
Enrollment: 7574 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | day 0
  Measured using the EQ-5D-5L score (EuroQoL score across 5 dimensions and 5 levels).
  EQ-5D-5L is measured on a scale between 0 and 1, where 0 is a state as bad as being dead, and 1 is full health.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Eggo, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- London School of Hygiene and Tropical Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The questionnaire data provided by participants will be made available to allow other researchers to benefit from this work in the future, and for a range of different studies and purposes. Opting-in to the study will require an affirmative response to agree to use of data in this way.
  After completion of the study, a pseudonymised copy of the data will be held according to NHS England retention policy, https://www.england.nhs.uk/contact-us/privacy-notice/how-we-use-your-information/covid-19-response/coronavirus-covid-19-research-platform/. Data access will be governed by London School of Hygiene and Tropical Medicine (LSHTM, data controller) and will require researchers to complete a data access form. This will be explained in all publications arising from the study.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The study protocol and informed consent form will be published in a study protocol paper in a peer reviewed medical journal.
  Analytic code will be shared as part of OpenSAFELY standards.

REFERENCES:
- [Derived] Herrett E, Tomlin K, Lin LY, Tomlinson LA, Jit M, Briggs A, Marks M, Sandmann F, Parry J, Bates C, Morley J, Bacon S, Butler-Cole B, Mahalingasivam V, Dennison A, Smith D, Gabriel E, Mehrkar A, Goldacre B, Smeeth L, Eggo RMM. Protocol for an OpenSAFELY cohort study collecting patient-reported outcome measures using the TPP Airmid smartphone application and linked big data to quantify the health and economic costs of long COVID (OpenPROMPT). BMJ Open. 2023 Feb 17;13(2):e071261. doi: 10.1136/bmjopen-2022-071261. PMID 36806073